CLINICAL TRIAL: NCT04007484
Title: The Effects of Hemoperfusion in Acute Type A Aortic Dissection Patients Undergoing Cardiopulmonary Bypass and Deep Hypothermic Circulatory Arrest: A Randomized, Controlled, Double-blinded Trial
Brief Title: Hemoperfusion in Acute Type A Aortic Dissection Patients Undergoing Aortic Arch Operation (HPAO)
Acronym: HPAO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP01PI
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2019-05

CONDITIONS: Acute Type A Aortic Dissection With Arch Involvement; Cardiopulmonary Bypass; Deep Hypothermic Circulatory Arrest
MeSH Terms: interventions — Hemoperfusion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HP+CPB/DHCA group (Experimental): For patients randomized into the intervention group, a hemoperfusion device will be connected in series to the extracorporeal circulation machine in advance to ensure that every single patient will undergo continuous hemoperfusion from the beginning to the end of CPB.
  Interventions: Device: Hemoperfusion
- CPB/DHCA group (No Intervention): For patients randomized into the CPB/DHCA group, no hemoperfusion device will be connect to the extracorporeal circulation machine. Patients will undergo CPB and DHCA without continuous hemoperfusion.

INTERVENTIONS:
Device: Hemoperfusion — Hemoperfusion is achieved by blood filtration with a hemoperfusion device. Specifically, the hemoperfusion device composed of multiple parallel resin cartridges is connected in parallel to the oxygenator and blood reservoir and perfused at a rate of 200-250ml/min. The purpose of hemoperfusion is to decrease inflammatory mediators produced during cardiopulmonary bypass through resin cartridges adsorption, such as cytokines, free hemoglobin and other toxins. The ultimate goal of hemoperfusion is to decrease postoperative complications, improve postoperative recovery, and eventually shorten the length of hospital stay.
  Arms: HP+CPB/DHCA group

SUMMARY:
This study is a single-center, randomized, controlled, double-blind clinical trial. The main purpose of this study is to evaluate if hemoperfusion is sufficient to improve the prognosis of acute type A aortic dissection patients undergoing cardiopulmonary bypass and deep hypothermia circulatory arrest.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 yr-75yr, regardless of gender
2. Patients with Acute type A aortic dissection and arch involvement (onset time ≤ 7 days)
3. Able to understand and sign the informed consent

Exclusion Criteria:

1. Unable to understand and sign the informed consent
2. BMI ≥ 40
3. Pregnant
4. Active hemorrhage or thrombocytopenic purpura
5. Previous history of liver diseasess, renal insufficiency or cerebrovascular diseases
6. Preoperative organ malperfusion
7. Previous history of cardiac surgeries
8. Oral anticoagulant or antiplatelet drugs within one week of disease onset
9. Hereditary connective tissue diseases such as Marfan syndrome, Ehlers-Danlos and Loeys-Dietz syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Composite major complications | up to 30 days
  Operative mortality, Secondary thoracotomy, New onset of postoperative renal failure requiring dialysis, Paraplegia, Stroke/cerebrovascular accidents, Low cardiac output syndrome, Reintubation, Severe liver dysfunction, ECMO support, Multiple organ dysfunction syndrome (MODS)

SECONDARY OUTCOMES:
Changes in the plasma levels of other inflammatory factors such as interleukin (IL)-6, IL-8, IL-10, IL-1β and TNF-α | up to 3 days
Changes of plasma MIF levels during the perioperative period | up to 3 days
Changes of plasma CRP levels during the perioperative period | up to 3 days
Total drainage within the first 24 hours of surgery | 24 hours
Incidence of postoperative acute kidney injury | up to 30 days
Incidence of postoperative respiratory failure | up to 30 days
Incidence of postoperative delirium | up to 30 days
Incidence of postoperative liver injury | up to 30 days
Incidence of postoperative myocardial infarction | up to 30 days
Changes of the plasma II, VII, IX, X, XI and XII levels during the perioperative period | up to 2 days
Changes of the plasma APTT, PT, FIB, FDP and DDi levels during the perioperative period | up to 3 days

OTHER OUTCOMES:
The need of vasoactive drugs | up to 30 days
  noradrenaline, epinephrine, dopamine and dobutamine
The volume of blood transfusion in ICU | up to 30 days
Length of ICU stay | up to 30 days
Length of postoperative stay | up to 30 days
Prolonged Postoperative Intubation | up to 30 days
  > 48h
Total hospital expenses | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Yang J, Ji D, Zhu YQ, Ren Y, Zhang X, Dai HY, Sun X, Zhou Y, Chen ZY, Li QG, Yao H. Hemoperfusion with HA380 in acute type A aortic dissection patients undergoing aortic arch operation (HPAO): a randomized, controlled, double-blind clinical trial. Trials. 2020 Nov 23;21(1):954. doi: 10.1186/s13063-020-04858-2. PMID 33228727